CLINICAL TRIAL: NCT00214500
Title: A Phase 2, Open-Label, Multicenter, 12-Week Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AT1001 in Patients With Fabry Disease
Brief Title: A Study of AT1001 (Migalastat Hydrochloride) in Participants With Fabry Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FAB-CL-201 (AA1565520); NCT00231036 (obsolete NCT alias)
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Results first posted 2018-09-07 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Fabry Disease
Keywords: Amicus Therapeutics; AT1001; Galafold; Migalastat; Substrate
MeSH Terms: conditions — Fabry Disease | interventions — migalastat; larazotide acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Migalastat (Experimental): Migalastat was administered orally during the 12-week treatment period and then during the optional 2 treatment extension periods.
  Treatment Period:
  * Migalastat 25 mg BID for Weeks 1 and 2 (Day 1 through the morning dose on Day 14).
  * Migalastat 100 mg BID for Weeks 3 and 4 (Day 15 through the morning dose on Day 28).
  * Migalastat 250 mg BID for Weeks 5 and 6 (Day 29 through the morning dose on Day 42).
  * Migalastat 25 mg BID for Weeks 6 to 12 (Days 43 to 84).
  Extension Period:
  * Migalastat 25 mg BID for Weeks 12 through 48.
  * Migalastat 50 mg QD for Weeks 48 through 96.
  Interventions: Drug: migalastat HCl

INTERVENTIONS:
Drug: migalastat HCl
  Other Names: AT1001; Galafold; migalastat

SUMMARY:
Study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of migalastat hydrochloride (HCl) (migalastat) in participants with Fabry disease.

DETAILED DESCRIPTION:
This was a Phase 2, open-label study in male participants with Fabry disease. All participants who met initial eligibility criteria underwent a 28-day screening period, including a 14-day run-in with migalastat (150 milligrams [mg] migalastat once a day [QD] from Days -28 to -15) to assess eligibility for entering the treatment period of the study. Participants who entered the treatment period were required to have α-galactosidase A (α-Gal A) activity responsive to migalastat.

Fifteen participants received at least 1 dose of study drug, however, 6 of these participants did not demonstrate α-Gal A activity responsive to migalastat and were thus screen failures (these participants are hereafter referred to as "dosed screen failures") due to not meeting all inclusion criteria for treatment. Therefore, 9 participants were enrolled into the treatment period (these participants are hereafter referred to as "eligible-enrolled").

Eligible-enrolled participants (those who satisfied the criteria for inclusion in the study) received escalating doses of migalastat twice a day (BID) for 6 weeks (Days 1 to 42), followed by 6 weeks at 1 dose level BID (Days 43 to 84) during the treatment period. Participants could then opt to participate in the extension period. The study consisted of 2 optional extension periods, the first through Week 48 and the second through Week 96. For participants who did not continue into the optional treatment extension, the study included a 2-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Males between 18 and 55 years of age (inclusive)
* Hemizygous for Fabry disease
* Had a confirmed diagnosis of Fabry disease with a documented missense gene mutation (individual or familial)
* Had enhanceable enzyme activity
* In the judgment of the investigator, were either able to safely suspend ERT throughout the study, or be ERT naive
* Agreed to be sexually abstinent or use a condom with spermicide when engaging in sexual activity during the course of the study and for a period of 30 days following completion of the study
* Were willing and able to sign an informed consent form

Exclusion Criteria:

* History of significant disease other than Fabry disease (for example, end-stage renal disease; Class III or IV heart disease [per the New York Heart Association classification]; current diagnosis of cancer, except for basal cell carcinoma of the skin; diabetes [unless hemoglobin A1c ≤8]; or neurological disease that would have impaired the participant's ability to participate in the study)
* History of organ transplant
* Serum creatinine >2 mg per deciliter on Day -2
* Screening 12-lead electrocardiogram demonstrating corrected QT interval >450 milliseconds prior to dosing
* Taking a medication prohibited by the protocol: Fabrazyme® (agalsidase beta), Replagal™ (agalsidase alfa), Glyset® (miglitol), Zavesca® (miglustat), or any experimental therapy for any indication
* Participated in a previous clinical trial in the last 30 days
* Any other condition, which, in the opinion of the investigator, would jeopardize the safety of the participant or impact the validity of the study results

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2006-01-02 (Actual); Primary Completion 2008-01-29 (Actual); Study Completion 2008-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Clinical Research, Study Director — Amicus Therapeutics
Locations (5):
- United States (5):
  - Los Angeles, California
  - Decatur, Georgia
  - Bethesda, Maryland
  - New York, New York
  - Houston, Texas

REFERENCES:
- [Derived] Benjamin ER, Della Valle MC, Wu X, Katz E, Pruthi F, Bond S, Bronfin B, Williams H, Yu J, Bichet DG, Germain DP, Giugliani R, Hughes D, Schiffmann R, Wilcox WR, Desnick RJ, Kirk J, Barth J, Barlow C, Valenzano KJ, Castelli J, Lockhart DJ. The validation of pharmacogenetics for the identification of Fabry patients to be treated with migalastat. Genet Med. 2017 Apr;19(4):430-438. doi: 10.1038/gim.2016.122. Epub 2016 Sep 22. PMID 27657681

RESULTS

PARTICIPANT FLOW:
Groups:
- Migalastat: Migalastat was administered orally during the 12-week treatment period and then during the optional 2 treatment extension periods.
  Treatment Period:
  * Migalastat 25 milligrams (mg) twice a day (BID) for Weeks 1 and 2 (Day 1 through the morning dose on Day 14).
  * Migalastat 100 mg BID for Weeks 3 and 4 (Day 15 through the morning dose on Day 28).
  * Migalastat 250 mg BID for Weeks 5 and 6 (Day 29 through the morning dose on Day 42).
  * Migalastat 25 mg BID for Weeks 6 to 12 (Days 43 to 84).
  Extension Period:
  * Migalastat 25 mg BID for Weeks 12 through 48.
  * Migalastat 50 mg once a day (QD) for Weeks 48 through 96.
Period: Treatment Period
Arm/Group | Migalastat
Started (6 additional participants were dosed screen failures and are not included) | 9 (All eligible-enrolled participants who received at least 1 dose of study drug)
Safety Population (All eligible-enrolled participants who received at least 1 dose of study drug) | 9
Pharmacokinetic (PK) Population (Received study drug and had at least 1 postbaseline PK parameter recorded) | 9
Pharmacodynamic (PD) Population (Received study drug on Day 1 and had a non-missing baseline and postbaseline PD parameter recorded) | 9
Completed | 8
Not Completed | 1
Not completed — Adverse Event | 1
Period: Extension Period
Arm/Group | Migalastat
Started | 8
Completed | 6
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Eligible-enrolled participants who received at least 1 dose of study drug. 6 participants were dosed screen failures, and were not included in safety, PK, or PD analyses.
Arm/Group | Migalastat
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (13.0)
Age, Customized [Count of Participants; unit: Participants] — 2 participants (aged 17 and 58) did not meet the age inclusion criterion but were granted approval by the Sponsor for enrollment before migalastat was administered.
  Participants
    17 years | 1
    18 to 55 years | 7
    58 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Number Of Participants Who Experienced Severe Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs were defined as any adverse event with start date on or after administration of study drug or pre-existing conditions that worsened on or after the start of the first study drug administration (on Day 1). A severe adverse event was defined as an adverse event that was incapacitating and required medical intervention. The number of participants who experienced one or more severe TEAEs after dosing on Day 1 through Week 96 is presented. A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Day 1 (after dosing) through Week 96
Population: Safety Population: all eligible-enrolled participants who received at least 1 dose of study drug. 6 participants were dosed screen failures, and were not included in the safety analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Migalastat
Number analyzed (Participants) | 9
Participants | 2

2. Secondary Outcome: PK: Area Under The Concentration Versus Time Curve (AUC) After Administration Of Migalastat
Description: The AUC from time zero to 12 hours (hr) postdose (AUC0-12) was evaluated in plasma following a single dose of migalastat 25, 100, and 250 mg on Days 1, 15, and 29, respectively. In addition, AUC0-12 was assessed following multiple doses (14 days) of migalastat 25, 100, and 250 mg on Days 14, 28, and 42, respectively.
Time Frame: 0 (predose), 0.5, 1, 2, 3, 4, 5, 6, 8, and 10 hr (postdose)
Population: PK Population: all eligible-enrolled participants who received study drug and had at least 1 postbaseline PK parameter recorded. One participant discontinued prior to receiving doses of migalastat 100 and 250 mg.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hr/milliliters (ng*hr/mL)
Groups:
- Migalastat 25 mg: Migalastat was administered orally. Migalastat 25 mg BID for Weeks 1 and 2 (Day 1 through the morning dose on Day 14).
- Migalastat 100 mg: Migalastat was administered orally. Migalastat 100 mg BID for Weeks 3 and 4 (Day 15 through the morning dose on Day 28).
- Migalastat 250 mg: Migalastat was administered orally. Migalastat 250 mg BID for Weeks 5 and 6 (Day 29 through the morning dose on Day 42).
Arm/Group | Migalastat 25 mg | Migalastat 100 mg | Migalastat 250 mg
Number analyzed (Participants) | 9 | 8 | 8
nanograms*hr/milliliters (ng*hr/mL)
  AUC0-12: Single Dose | 1052.96 (29.9) | 4217.95 (32.0) | 10880.66 (32.4)
  AUC0-12: Multiple Dose | 1360.69 (32.9) | 5643.50 (25.3) | 12244.47 (26.0)

3. Secondary Outcome: α-Galactosidase A (α-Gal A) Activity In Leukocytes At Baseline, Week 12, And Week 96
Description: Leukocytes were isolated from whole blood and lysed, and α-Gal A activity was measured using a validated fluorometric assay, with catalysis to fluorescent 4-methylumbelliferone (4-MU) as the activity measure. The activity values obtained were normalized to protein (measured using a colorimetric assay) and reported as enzyme activity (nanomole [nmol] 4-MU/hr) per mg of protein. On Day 1 of the first visit and at every visit thereafter, the samples were collected prior to dosing with migalastat. α-Gal A activity in leukocytes are presented by individual participants.
Time Frame: Baseline, Week 12 (end of treatment period), Week 96 (end of extension period)
Population: PD Population: all eligible-enrolled participants who received at least 1 dose of study drug on Day 1, and who had a non-missing baseline and at least 1 non-missing postbaseline PD parameter recorded. Participants who discontinued prior to the specified time point were not analyzed because no data were available.
Measure: Number; unit: nmol 4-MU/hr/mg protein
Arm/Group | Migalastat
Number analyzed (Participants) | 9
nmol 4-MU/hr/mg protein
  Participant 1: Baseline: number analyzed (Participants) | 1
  Participant 1: Baseline | 5.2
  Participant 1: Week 12: number analyzed (Participants) | 1
  Participant 1: Week 12 | 17.4
  Participant 1: Week 96: number analyzed (Participants) | 1
  Participant 1: Week 96 | 20.3
  Participant 2: Baseline: number analyzed (Participants) | 1
  Participant 2: Baseline | 4.7
  Participant 2: Week 12: number analyzed (Participants) | 1
  Participant 2: Week 12 | 24.6
  Participant 2: Week 96: number analyzed (Participants) | 1
  Participant 2: Week 96 | 22.8
  Participant 3: Baseline: number analyzed (Participants) | 1
  Participant 3: Baseline | 6.6
  Participant 3: Week 12: number analyzed (Participants) | 1
  Participant 3: Week 12 | 24.6
  Participant 3: Week 96: number analyzed (Participants) | 1
  Participant 3: Week 96 | 20.3
  Participant 4: Baseline: number analyzed (Participants) | 1
  Participant 4: Baseline | 1.0
  Participant 4: Week 12: number analyzed (Participants) | 1
  Participant 4: Week 12 | 14.8
  Participant 4: Week 96: number analyzed (Participants) | 1
  Participant 4: Week 96 | 12.8
  Participant 5: Baseline: number analyzed (Participants) | 1
  Participant 5: Baseline | 10.7
  Participant 5: Week 12: number analyzed (Participants) | 0
  Participant 5: Week 96: number analyzed (Participants) | 0
  Participant 6: Baseline: number analyzed (Participants) | 1
  Participant 6: Baseline | 0.9
  Participant 6: Week 12: number analyzed (Participants) | 1
  Participant 6: Week 12 | 3.9
  Participant 6: Week 96: number analyzed (Participants) | 1
  Participant 6: Week 96 | 1.9
  Participant 7: Baseline: number analyzed (Participants) | 1
  Participant 7: Baseline | 0.0
  Participant 7: Week 12: number analyzed (Participants) | 1
  Participant 7: Week 12 | 0.4
  Participant 7: Week 96: number analyzed (Participants) | 0
  Participant 8: Baseline: number analyzed (Participants) | 1
  Participant 8: Baseline | 0.1
  Participant 8: Week 12: number analyzed (Participants) | 1
  Participant 8: Week 12 | 0.9
  Participant 8: Week 96: number analyzed (Participants) | 0
  Participant 9: Baseline: number analyzed (Participants) | 1
  Participant 9: Baseline | 0.2
  Participant 9: Week 12: number analyzed (Participants) | 1
  Participant 9: Week 12 | 0.3
  Participant 9: Week 96: number analyzed (Participants) | 1
  Participant 9: Week 96 | 0.2

ADVERSE EVENTS:
Time Frame: Day 1 after dosing through Week 96 (end of extension period)
Arm/Group | Migalastat
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 9/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Migalastat (N=9)
Abdominal pain upper (Gastrointestinal disorders) | 2
Angiokeratoma (Skin and subcutaneous tissue disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bipolar disorder (Psychiatric disorders) | 1
Blood bilirubin increased (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Blood glucose increased (Investigations) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Deafness (Ear and labyrinth disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Fatigue (General disorders) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Giardiasis (Infections and infestations) | 1
Gingival pain (Gastrointestinal disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Headache (Nervous system disorders) | 5
Hunger (General disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Influenza like illness (General disorders) | 1
Insomnia (Psychiatric disorders) | 2
Libido decreased (Psychiatric disorders) | 1
Micturition urgency (Renal and urinary disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nasopharyngitis (Infections and infestations) | 1
Nausea (Gastrointestinal disorders) | 4
Odynophagia (Gastrointestinal disorders) | 1
Oedema peripheral (General disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Pain (General disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Pyrexia (General disorders) | 1
Respiratory tract infection (Infections and infestations) | 1
Respiratory tract irritation (Respiratory, thoracic and mediastinal disorders) | 1
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1
Thirst (General disorders) | 1
Tinea versicolour (Infections and infestations) | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Vertigo (Ear and labyrinth disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator can only publish the results from this trial provided they supply the sponsor (or authorized entity) a copy of any proposed publication for review. If requested, the investigator will remove information deemed confidential or proprietary by the sponsor and will withhold publication for an additional period of time to allow the sponsor to take appropriate measures to establish and preserve its proprietary rights.